CLINICAL TRIAL: NCT01877434
Title: The TESS Reverse Shoulder Arthroplasty: Effect of Arm Lengthening and Early Scapular Notching at Three Years Follow-up
Brief Title: Reversed TESS Shoulder Artroplasty
Acronym: RTESS
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Principal Investigator, Lennart Bråbäck, Consultat medical doctor, Sundsvall Hospital
Other Study IDs: 2012-201-31M
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Humerus Fracture; Degenerative Shoulder Pain; Degenerative Supraspinatus Rupture
Keywords: Reversed shoulder arthroplasty; Treatment; TESS
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Reversed TESS: Patient undergone reversed shoulder arthroplasty
  Interventions: Procedure: Reversed shoulder arthroplasty

INTERVENTIONS:
Procedure: Reversed shoulder arthroplasty

SUMMARY:
Reverse total shoulder arthroplasty (RSA) is a accepted treatment for different shoulder diseases with improved functional outcome. This study has evaluated patients operated with reversed shoulder arthroplasty after 1,5-3 years postoperatively with patient reported outcome, clinical and radiological examination, complication and reoperations. The radiologic phenomenom and clinical impact of scapular notching (SN) and arm length difference has been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Operated with a reversed TESS total shoulder arthroplasty at Sundsvall hospital.

Exclusion Criteria:

* Do not give informed consent
* Do not attend follow-up

Ages: 60 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergone reversed shoulder arthroplasty at Sundsvall hospital, Sweden between 2007-2012
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2012-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Patient reported outcome measurement Quick-DASH | 2007-2013

SECONDARY OUTCOMES:
Range of movement | 2007-2013
Quality of life EQ5-D | 2007-2013

OTHER OUTCOMES:
Arm lenght difference | 2007-2013
  Impact on arm lenght difference on patient reported outcome evaluated with Quick-DASH

CONTACTS AND LOCATIONS:
Locations (1):
- Institution of surgical and operative sciences, Umeå University, Sundsvall, Västernorrland Län, Sweden